CLINICAL TRIAL: NCT01220778
Title: Effects of Physical Activity During Pregnancy on the Newborn's Cognitive Function, the Healthy Mom, Bright Child Randomized Trial
Brief Title: Effects of Physical Activity During Pregnancy on the Newborn's Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Allocation: Randomized | Model: Parallel
Other Study IDs: CERSS-2010-951-P
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-09

CONDITIONS: Pregnancy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise

SUMMARY:
Background: It is now generally accepted that an active lifestyle is beneficial for cognition, but can these benefits be transmitted for the active pregnant woman to her unborn child? This has been demonstrated in rats where the pups born of mothers who exercised during pregnancy had increased hippocampal neurogenesis and better memory and learning capabilities. Human studies tend to confirm this by looking at behavioral results, ie. better orientation and state regulation skills in newborns. The aim of the present study is to verify this on the electrophysiological level and to determine the effects of an active lifestyle during pregnancy on the newborn's brain development.

Methods: 60 pregnant women will be included in a randomized controlled trial. The exercise group will be asked to exercise a minimum of 20 minutes, 3 times per week, at a minimal intensity of 55% of their maximal aerobic capacity. The control group will not be given exercise counselling. Newborns' brain activity will be recorded using electroencephalography (EEG) 10 days post partum. The primary outcome measure will be the amplitude and latency of the mismatch negativity (MMN), a component of the auditory event-related potential (ERP) that can be used to investigate the auditory sensory memory.

ELIGIBILITY:
Inclusion Criteria:

* First trimester of pregnancy
* 20 to 35 years of age
* Pre-pregnancy BMI between 18 and 25
* Primipara
* Without any known health issues
* Use of folic acid

Exclusion Criteria:

* Use of alcohol, cigarettes or illegal drugs
* Pregnancy complications
* Unable or unwilling to breastfeed
* Excessive or insufficient weight gain

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult

PRIMARY OUTCOMES:
Mismatch negativity

CONTACTS AND LOCATIONS:
Overall Officials: Elise L.LeMoyne, Principal Investigator — Université de Montréal
Locations (1):
- Cepsum, Montreal, Quebec, Canada

REFERENCES:
- [Derived] LeMoyne EL, Curnier D, St-Jacques S, Ellemberg D. The effects of exercise during pregnancy on the newborn's brain: study protocol for a randomized controlled trial. Trials. 2012 May 29;13:68. doi: 10.1186/1745-6215-13-68. PMID 22643160